CLINICAL TRIAL: NCT04159207
Title: A Longitudinal Study of Inflammatory Pathways in Depression
Status: Completed | Type: Observational
Sponsor: Van Andel Research Institute (Other)
Collaborators: Pine Rest Christian Mental Health Services (Other); Columbia University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lena Brundin, Associate Professor, Van Andel Research Institute
Other Study IDs: 19010; 1R01MH118211-01A1 (NIH)
Record Dates: First submitted 2019-09-30; First posted 2019-11-12 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder; Suicide, Attempted
Keywords: Depression; Suicide; Inflammation; Kynurenine; Cytokine
MeSH Terms: conditions — Depressive Disorder, Major; Suicide, Attempted; Depression; Suicide; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- A Longitudinal Study of Inflammatory Pathways in Depression: We target to recruit 80 patients with Major Depression Disorder diagnosis and 80 patients with Major Depression Disorder with suicidal behavior.

SUMMARY:
Suicide accounts for at least 1 million deaths globally each year. This is likely a significant underestimate, because suicide is under-reported in many countries. In the US, over 42,000 people die from suicide annually. Despite increased focus on identification and treatment, the rate of suicide has increased steadily over the past 15 years.

Our project aims both to improve our understanding of factors that increase the risk for suicide by comparing blood biomarkers associated with inflammation in patients with depression without suicidal behavior and patients with depression and suicidal behavior. The 160 individuals in this study will be followed with psychiatric assessments and blood samples at repeated time points over one year.

DETAILED DESCRIPTION:
Suicide is a leading cause of death in the US, and its rate continues to increase. Most individuals who die by suicide are in contact with health care, but clinical risk assessment is challenging. Inflammatory biomarkers have tentatively been linked to suicide. However, longitudinal studies establishing their accuracy in tracking suicidal behavior and critical symptoms are lacking. This study is a longitudinal study, with 1,280 total assessments planned, measuring suicidal ideation and behavior, associated clinical symptoms and blood biomarkers of inflammation.

Our overriding aim is to identify a set of biomarkers that distinguish patients with suicidal behavior from depressive patients without suicidal behavior. Further, the investigators intend to define biomarkers that are elevated during active suicidal behavior (at- risk periods) within the same patients (longitudinally).

Our working model is that inflammation (via pro-inflammatory cytokines) induces the kynurenine pathway, leading to an increased production of neurotoxic kynurenine metabolites (i.e., the NMDA-receptor agonist quinolinic acid, or others), which trigger suicidal behavior. The Investigators predict that immunomodulatory cells and molecules, including cytokines and kynurenine metabolites in plasma, may constitute biomarkers of suicidal behavior. The Investigators also predict that elevated inflammatory markers in suicidal individuals will be associated with epigenetic changes, regulating the expression of kynurenine enzymes in blood cells.

Aims:

1. Establish biomarkers that indicate risk for active suicidal behavior;
2. Determine epigenetic markers in the blood of patients with suicidal behavior.

In Aim 1, the investigators will enroll patients with Major Depressive Disorder (MDD) and active suicidal behavior (planning or attempts), and MDD patients without current or past suicidal behavior. Each subject will be assessed at eight time-points over one year. The Investigators will measure interleukins and acute phase reactants as well as tryptophan, serotonin and metabolites of the kynurenine pathway in peripheral blood.

For aim 2, the investigators will perform whole-genome methylation analysis using Illumina EPIC arrays, followed by gene pathway analyses, in blood of the enrolled patients.

Our project will aid the implementation of biomarkers in clinical care for patients with suicide risk, in order to enable intensified intervention during critical time-points. The biological insight obtained here can guide therapeutic development specifically targeting suicidality, with the ultimate goal of reducing suicide numbers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 years and older will be included in the study.
* 80 who are diagnosed with MDD by SCID but do not endorse current or past suicidal behaviors.
* 80 who are diagnosed with MDD by SCID and endorse current suicidal behavior as defined by C-SSRS (preparatory acts, aborted or interrupted attempts, as well as completed attempts).
* English speaking.
* Willing and able to take part of the different steps in the study, including follow-up interviews and blood draws.

Exclusion Criteria:

* Vulnerable populations (e.g. incarcerated individuals).
* Subjects with dementia or otherwise cognitively impaired subjects with difficulty understanding the study procedures.
* Patients with a primary psychiatric diagnosis other than MDD.
* Patients with an active somatic disorder primarily involving the immune system (autoimmune diseases such as Crohns disease, multiple sclerosis, or rheumatoid arthritis; or hematological diseases such as lymphoma or leukemia).
* Patients on chronic and systemic immunomodulatory treatment. Examples are patients with a liver- or kidney transplant or medications used for disorders involving the immune system, as mentioned above. Examples of immunomodulatory treatments are cyclosporin, azathioprine, infliximab, corticosteroid treatment.
* Patients undergoing active treatment for any form of cancer (chemotherapy or immunomodulatory treatments).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are above age of 18, have a Major Depressive Disorder diagnosis and no ongoing immune disorders.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Suicidal behavior of participants | One year.
  The presence of suicidal behavior over one year will be classified as yes/no as the primary outcome measure. The Identification of participants with suicidal behavior at each study time point will be achieved by assessment using the Columbia Suicide Severity Rating Scale (C-SSRS) regarding attempt, interrupted or aborted attempt, or preparatory acts over the past 7 days.
Establish metabolic biomarkers that indicate risk for suicidal behavior | One year.
  Evaluate if metabolic biomarkers are predictive of suicidal behavior (planning, attempting) among patients with depression. Metabolites will be measured by high-pressure liquid chromatography, ultra-high performace liquid-chromatography and gas-chromatography mass-spectrometry). The main metabolite biomarker outcomes are quinolinic, kynurenic and picolinic acids as well as 3-HK and kynurenine (nM).
Establish inflammatory biomarkers that indicate risk for suicidal behavior | One year.
  Evaluate if inflammatory biomarkers are predictive of suicidal behavior (planning, attempting) among patients with depression. Inflammatory markers will be measured using high-sensitivity ELISAs, Mesoscale platform or Luminex platforms. The main cytokine outcomes are TNF-alpha and IL-6 (pg/ml).
Determine epigenetic marks in blood cells from patients with suicidal behavior | One year.
  DNA methylation will be measured by Illumina Infinum methylationEPIC BeadChip microarrays, and compacted between patients with suicidal behavior and patients without suicidal behavior.
Functional validation of the significant methylation changes | One year.
  mRNA will be quantified by qPCR in the same peripheral blood samples as used for the EPIC array for functional validation of the significant methylation changes.

CONTACTS AND LOCATIONS:
Overall Officials: Lena C Brundin, M.D.; Ph.D., Principal Investigator — Van Andel Research Institute; Eric Achtyes, M.D., Principal Investigator — Pine Rest Christian Mental Health Services; Joseph Mann, M.D., Principal Investigator — Columbia University Health Sciences
Locations (1):
- Pine Rest Christian Mental Health Services, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Center for Disease Control and Prevention. Preventing Suicide. 2018.
- [Background] Shepard DS, Gurewich D, Lwin AK, Reed GA Jr, Silverman MM. Suicide and Suicidal Attempts in the United States: Costs and Policy Implications. Suicide Life Threat Behav. 2016 Jun;46(3):352-62. doi: 10.1111/sltb.12225. Epub 2015 Oct 29. PMID 26511788
- [Background] Curtin SC, Warner M, Hedegaard H. Increase in Suicide in the United States, 1999-2014. NCHS Data Brief. 2016 Apr;(241):1-8. PMID 27111185
- [Background] Lutz PE, Mechawar N, Turecki G. Neuropathology of suicide: recent findings and future directions. Mol Psychiatry. 2017 Oct;22(10):1395-1412. doi: 10.1038/mp.2017.141. Epub 2017 Jul 11. PMID 28696430
- [Background] Roy B, Dwivedi Y. Understanding epigenetic architecture of suicide neurobiology: A critical perspective. Neurosci Biobehav Rev. 2017 Jan;72:10-27. doi: 10.1016/j.neubiorev.2016.10.031. Epub 2016 Nov 9. PMID 27836463
- [Background] Black C, Miller BJ. Meta-Analysis of Cytokines and Chemokines in Suicidality: Distinguishing Suicidal Versus Nonsuicidal Patients. Biol Psychiatry. 2015 Jul 1;78(1):28-37. doi: 10.1016/j.biopsych.2014.10.014. Epub 2014 Oct 30. PMID 25541493
- [Background] Bryleva EY, Brundin L. Suicidality and Activation of the Kynurenine Pathway of Tryptophan Metabolism. Curr Top Behav Neurosci. 2017;31:269-284. doi: 10.1007/7854_2016_5. PMID 27221623
- [Background] Gananca L, Oquendo MA, Tyrka AR, Cisneros-Trujillo S, Mann JJ, Sublette ME. The role of cytokines in the pathophysiology of suicidal behavior. Psychoneuroendocrinology. 2016 Jan;63:296-310. doi: 10.1016/j.psyneuen.2015.10.008. Epub 2015 Oct 19. PMID 26546783
- [Background] Miyaoka H, Otsubo T, Kamijima K, Ishii M, Onuki M, Mitamura K. Depression from interferon therapy in patients with hepatitis C. Am J Psychiatry. 1999 Jul;156(7):1120. doi: 10.1176/ajp.156.7.1120. No abstract available. PMID 10401474
- [Background] Lucaciu LA, Dumitrascu DL. Depression and suicide ideation in chronic hepatitis C patients untreated and treated with interferon: prevalence, prevention, and treatment. Ann Gastroenterol. 2015 Oct-Dec;28(4):440-7. PMID 26424594
- [Background] Yirmiya R, Pollak Y, Morag M, Reichenberg A, Barak O, Avitsur R, Shavit Y, Ovadia H, Weidenfeld J, Morag A, Newman ME, Pollmacher T. Illness, cytokines, and depression. Ann N Y Acad Sci. 2000;917:478-87. doi: 10.1111/j.1749-6632.2000.tb05412.x. PMID 11268375
- [Background] Yirmiya R. Endotoxin produces a depressive-like episode in rats. Brain Res. 1996 Mar 4;711(1-2):163-74. doi: 10.1016/0006-8993(95)01415-2. PMID 8680860
- [Background] O'Connor JC, Lawson MA, Andre C, Moreau M, Lestage J, Castanon N, Kelley KW, Dantzer R. Lipopolysaccharide-induced depressive-like behavior is mediated by indoleamine 2,3-dioxygenase activation in mice. Mol Psychiatry. 2009 May;14(5):511-22. doi: 10.1038/sj.mp.4002148. Epub 2008 Jan 15. PMID 18195714
- [Background] Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biol Psychiatry. 2010 Mar 1;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. Epub 2009 Dec 16. PMID 20015486
- [Background] Dahl J, Ormstad H, Aass HC, Malt UF, Bendz LT, Sandvik L, Brundin L, Andreassen OA. The plasma levels of various cytokines are increased during ongoing depression and are reduced to normal levels after recovery. Psychoneuroendocrinology. 2014 Jul;45:77-86. doi: 10.1016/j.psyneuen.2014.03.019. Epub 2014 Apr 6. PMID 24845179
- [Background] Tonelli LH, Stiller J, Rujescu D, Giegling I, Schneider B, Maurer K, Schnabel A, Moller HJ, Chen HH, Postolache TT. Elevated cytokine expression in the orbitofrontal cortex of victims of suicide. Acta Psychiatr Scand. 2008 Mar;117(3):198-206. doi: 10.1111/j.1600-0447.2007.01128.x. Epub 2007 Dec 13. PMID 18081924
- [Background] Steiner J, Bielau H, Brisch R, Danos P, Ullrich O, Mawrin C, Bernstein HG, Bogerts B. Immunological aspects in the neurobiology of suicide: elevated microglial density in schizophrenia and depression is associated with suicide. J Psychiatr Res. 2008 Jan;42(2):151-7. doi: 10.1016/j.jpsychires.2006.10.013. Epub 2006 Dec 15. PMID 17174336
- [Background] Pandey GN, Rizavi HS, Ren X, Fareed J, Hoppensteadt DA, Roberts RC, Conley RR, Dwivedi Y. Proinflammatory cytokines in the prefrontal cortex of teenage suicide victims. J Psychiatr Res. 2012 Jan;46(1):57-63. doi: 10.1016/j.jpsychires.2011.08.006. Epub 2011 Sep 8. PMID 21906753
- [Background] Torres-Platas SG, Cruceanu C, Chen GG, Turecki G, Mechawar N. Evidence for increased microglial priming and macrophage recruitment in the dorsal anterior cingulate white matter of depressed suicides. Brain Behav Immun. 2014 Nov;42:50-9. doi: 10.1016/j.bbi.2014.05.007. Epub 2014 May 20. PMID 24858659
- [Background] Holmes SE, Hinz R, Conen S, Gregory CJ, Matthews JC, Anton-Rodriguez JM, Gerhard A, Talbot PS. Elevated Translocator Protein in Anterior Cingulate in Major Depression and a Role for Inflammation in Suicidal Thinking: A Positron Emission Tomography Study. Biol Psychiatry. 2018 Jan 1;83(1):61-69. doi: 10.1016/j.biopsych.2017.08.005. Epub 2017 Aug 12. PMID 28939116
- [Background] O'Donovan A, Rush G, Hoatam G, Hughes BM, McCrohan A, Kelleher C, O'Farrelly C, Malone KM. Suicidal ideation is associated with elevated inflammation in patients with major depressive disorder. Depress Anxiety. 2013 Apr;30(4):307-14. doi: 10.1002/da.22087. Epub 2013 Mar 15. PMID 23504697
- [Background] Janelidze S, Mattei D, Westrin A, Traskman-Bendz L, Brundin L. Cytokine levels in the blood may distinguish suicide attempters from depressed patients. Brain Behav Immun. 2011 Feb;25(2):335-9. doi: 10.1016/j.bbi.2010.10.010. Epub 2010 Oct 15. PMID 20951793
- [Background] Dantzer R, O'Connor JC, Freund GG, Johnson RW, Kelley KW. From inflammation to sickness and depression: when the immune system subjugates the brain. Nat Rev Neurosci. 2008 Jan;9(1):46-56. doi: 10.1038/nrn2297. PMID 18073775
- [Background] Bayard-Burfield L, Alling C, Blennow K, Jonsson S, Traskman-Bendz L. Impairment of the blood-CSF barrier in suicide attempters. Eur Neuropsychopharmacol. 1996 Aug;6(3):195-9. doi: 10.1016/0924-977x(96)00020-x. PMID 8880079
- [Background] Falcone T, Fazio V, Lee C, Simon B, Franco K, Marchi N, Janigro D. Serum S100B: a potential biomarker for suicidality in adolescents? PLoS One. 2010 Jun 14;5(6):e11089. doi: 10.1371/journal.pone.0011089. PMID 20559426
- [Background] Ventorp F, Barzilay R, Erhardt S, Samuelsson M, Traskman-Bendz L, Janelidze S, Weizman A, Offen D, Brundin L. The CD44 ligand hyaluronic acid is elevated in the cerebrospinal fluid of suicide attempters and is associated with increased blood-brain barrier permeability. J Affect Disord. 2016 Mar 15;193:349-54. doi: 10.1016/j.jad.2015.12.069. Epub 2016 Jan 6. PMID 26796235
- [Background] Dantzer R, Kelley KW. Stress and immunity: an integrated view of relationships between the brain and the immune system. Life Sci. 1989;44(26):1995-2008. doi: 10.1016/0024-3205(89)90345-7. PMID 2568569
- [Background] McGirr A, Renaud J, Bureau A, Seguin M, Lesage A, Turecki G. Impulsive-aggressive behaviours and completed suicide across the life cycle: a predisposition for younger age of suicide. Psychol Med. 2008 Mar;38(3):407-17. doi: 10.1017/S0033291707001419. Epub 2007 Sep 6. PMID 17803833
- [Background] Isung J, Aeinehband S, Mobarrez F, Nordstrom P, Runeson B, Asberg M, Piehl F, Jokinen J. High interleukin-6 and impulsivity: determining the role of endophenotypes in attempted suicide. Transl Psychiatry. 2014 Oct 21;4(10):e470. doi: 10.1038/tp.2014.113. PMID 25335166
- [Background] Coccaro EF, Lee R, Coussons-Read M. Elevated plasma inflammatory markers in individuals with intermittent explosive disorder and correlation with aggression in humans. JAMA Psychiatry. 2014 Feb;71(2):158-65. doi: 10.1001/jamapsychiatry.2013.3297. PMID 24352431
- [Background] Schwieler L, Larsson MK, Skogh E, Kegel ME, Orhan F, Abdelmoaty S, Finn A, Bhat M, Samuelsson M, Lundberg K, Dahl ML, Sellgren C, Schuppe-Koistinen I, Svensson C, Erhardt S, Engberg G. Increased levels of IL-6 in the cerebrospinal fluid of patients with chronic schizophrenia--significance for activation of the kynurenine pathway. J Psychiatry Neurosci. 2015 Mar;40(2):126-33. doi: 10.1503/jpn.140126. PMID 25455350
- [Background] Tavares RG, Tasca CI, Santos CE, Alves LB, Porciuncula LO, Emanuelli T, Souza DO. Quinolinic acid stimulates synaptosomal glutamate release and inhibits glutamate uptake into astrocytes. Neurochem Int. 2002 Jun;40(7):621-7. doi: 10.1016/s0197-0186(01)00133-4. PMID 11900857
- [Background] Stone TW. Neuropharmacology of quinolinic and kynurenic acids. Pharmacol Rev. 1993 Sep;45(3):309-79. PMID 8248282
- [Background] Hilmas C, Pereira EF, Alkondon M, Rassoulpour A, Schwarcz R, Albuquerque EX. The brain metabolite kynurenic acid inhibits alpha7 nicotinic receptor activity and increases non-alpha7 nicotinic receptor expression: physiopathological implications. J Neurosci. 2001 Oct 1;21(19):7463-73. doi: 10.1523/JNEUROSCI.21-19-07463.2001. PMID 11567036
- [Background] Sublette ME, Galfalvy HC, Fuchs D, Lapidus M, Grunebaum MF, Oquendo MA, Mann JJ, Postolache TT. Plasma kynurenine levels are elevated in suicide attempters with major depressive disorder. Brain Behav Immun. 2011 Aug;25(6):1272-8. doi: 10.1016/j.bbi.2011.05.002. Epub 2011 May 14. PMID 21605657
- [Background] Bradley KA, Case JA, Khan O, Ricart T, Hanna A, Alonso CM, Gabbay V. The role of the kynurenine pathway in suicidality in adolescent major depressive disorder. Psychiatry Res. 2015 Jun 30;227(2-3):206-12. doi: 10.1016/j.psychres.2015.03.031. Epub 2015 Apr 1. PMID 25865484